CLINICAL TRIAL: NCT06819475
Title: Imaging Skeletal Muscle Mitochondrial OXPHOS Activity In Acute Lymphoblastic Leukemia Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: MMICCS; NCI-2024-09771 (Other: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2025-01-08; First posted 2025-02-11 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Childhood Cancer; Muscle Weakness
Keywords: Survivor; Acute Lymphoblastic Leukemia; Adult; ALL; Healthy Volunteer
MeSH Terms: conditions — Neoplasms; Muscle Weakness; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Magnetic Resonance Imaging; Positron-Emission Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Survivors (Experimental): Adult survivor of acute lymphoblastic leukemia (ALL) enrolled in St. Jude Life Cohort (SJLIFE).
  Interventions: Diagnostic Test: Magnetic Resonance Imaging; Diagnostic Test: Magnetic Resonance Spectroscopy; Other: Physical function assessment; Other: Peripheral blood sample; Other: Skeletal muscle biopsy; Diagnostic Test: Muscle Ultrasound
- Control (Experimental): Control participants are not a close relative of someone who has received treatment for childhood cancer or a similar illness; age/sex-matched healthy volunteers and recruited from SJLIFE Control cohort and may be recruited from new SJLIFE Controls.
  Interventions: Diagnostic Test: Magnetic Resonance Imaging; Diagnostic Test: Magnetic Resonance Spectroscopy; Other: Physical function assessment; Other: Peripheral blood sample; Other: Skeletal muscle biopsy; Diagnostic Test: Muscle Ultrasound

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging — Non-invasive MRI will be used to measure the major muscle groups in the calf muscle mtOXPHOS in childhood survivors of Acute Lymphoblastic Leukemia (ALL) in SJLIFE cohort and healthy controls and measure how muscle mitochondria produce energy to function.
  Other Names: MRI
Diagnostic Test: Magnetic Resonance Spectroscopy — Non-invasive MRS will be used to measure the major muscle groups in the calf muscle mtOXPHOS in childhood survivors of Acute Lymphoblastic Leukemia (ALL) in SJLIFE cohort and healthy controls and measure how muscle mitochondria produce energy to function.
  Other Names: MRS
Other: Physical function assessment — As part of the SJLIFE visit in the Human Performance Lab, the participant's physical health will be assessed by testing muscle strength, physical function, and lean muscle mass.
Other: Peripheral blood sample — Peripheral blood sample will be used to evaluate muscle morphology, mitochondrial health and epigenetic differences in the muscles of survivors and age/sex-matched healthy controls.
Other: Skeletal muscle biopsy — Muscle biopsy will be used to evaluate muscle morphology, mitochondrial health and epigenetic differences in muscles of survivors and age/sex-matched healthy controls.
Diagnostic Test: Muscle Ultrasound — Bilateral quadriceps and calf muscle ultrasound will be used to measure muscle volume by calculating the cross-sectional area using the Cavalieri method.

SUMMARY:
The participants are being asked to take part in this trial, because the participant is a survivor of childhood cancer or agreed to be part of a volunteer group to understand the relation between cancer and cancer treatment and muscle weakness in survivors of Acute Lymphoblastic Leukemia (ALL). ALL is cancer of the blood and bone marrow.

Primary Objective

• To compare muscle mtOXPHOS activity and satellite cell content among ALL survivors and controls.

Secondary Objective

* To evaluate the association between muscle mtOXPHOS, muscle satellite cell content and physical performance in ALL survivors.
* To evaluate the association of muscle morphology and epigenetics with muscle mtOXPHOS in ALL survivors.

DETAILED DESCRIPTION:
This study hypothesizes that sarcopenia (low lean mass and muscle weakness), the central components of frailty, result from cancer- and or treatment-related impairment of cellular function within skeletal myocytes. Impaired mitochondrial oxidative phosphorylation (mtOXPHOS) is a hallmark of aging and implicated in skeletal muscle (muscle) weakness and lowered physical performance with normal aging. There is a lack of understanding of how the dysfunctional mitochondrial capacity affects the individual muscle groups in the lower extremities of the survivors.

This pilot study will explore the feasibility of non-invasive metabolic imaging to measure the major muscle groups in the calf muscle mtOXPHOS in childhood survivors of Acute Lymphoblastic Leukemia (ALL) in SJLIFE cohort by incorporating magnetic resonance imaging (MRI) and magnetic resonance spectroscopy (MRS) in survivors and age/sex-matched healthy volunteers (Controls). Control participants will be recruited from SJLIFE control cohort and may be recruited from new SJLIFE controls; The MRI/MRS findings will be correlated with clinically ascertained muscle phenotype; and will explore and describe differences in muscle morphology, epigenetics, mtDNA-CN between survivors and controls using peripheral blood and muscle biopsies, and their association with MRI/MRS findings.

Survivor and Control participants will be asked to have two MRI sessions; a physical function, and a muscle ultrasound assessment done during SJLIFE Human Performance Lab (HPL). Participants will be asked to give a peripheral blood sample and muscle sample. MR imaging will be performed in two appointments.

ELIGIBILITY:
Inclusion Criteria:

* Survivor- or Control-Participant is age 18 years old or older at time of consent and enrolled in SJLIFE.
* Survivor- Participant is childhood ALL survivor
* Survivor- or Control Participant has low muscle mass as defined by relative lean mass z-score of less than or equal to -0.5 SD (lean mass divided by height in meters squared).
* Survivor- or Control-Participant is able and willing to give informed consent

Exclusion Criteria:

* Survivor-Participant has history of cranial radiation.
* Survivor- or Control-Participant has implanted medical devices or metal that would interfere with MRI or MRS
* Female Survivor- or Control-Participant is pregnant.
* Survivor- or Control-Participant is taking anticoagulants (e.g. aspirin, apixaban, coumadin, edoxaban, rivaroxaban)
* Survivor- or Control-Participant weighs more than 300 pounds.
* Survivor- or Control-Participant is allergic to local anesthetic (i.e., lidocaine, bupivacaine).
* Survivor- or Control-Participant cannot lie flat on his/her back for 90 minutes or longer
* Survivor- or Control-Participant has a current history of peripheral motor neuropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
To explore feasibility of MRI/MRS to measure OXPHOS capacity | Baseline
  Multimodal MR imaging will be performed in two appointments. The first appointment will consist of Part 1 (approximately 1 hour) and Part 2 (approximately 30 minutes). There will be a 5-10 minute break between the two parts. The second appointment will consist of Part 1 (approximately 1 hour).
To explore feasibility of 31P-MRS to measure OXPHOS capacity | Baseline
  This will be performed with a 7-cm diameter 1H/31P dual-tuned surface/volume coil using an unlocalized free induction decay (FID) sequence: number of points = 512, averages = 2-5, and TR = 2.4-5 seconds, with 4 dummy scans. TPCr is determined by fitting the signal intensity of PCr following plantar flexion exercise to a mono-exponential function. Additionally, we will acquire a steady state 31P-MR spectra for phosphorylated metabolite quantification (sec).
To explore feasibility of 1H-MRS to measure OXPHOS capacity | Baseline
  This will be performed on a Siemens 3T scanner using Point RESolved Spectroscopy (PRESS) 31 sequence. A water-suppressed 1H MR spectrum will be acquired from a voxel positioned in gastrocnemius and soleus muscles. 1H MRS data will be processed using LCModel providing the metabolite levels (mM).
To explore feasibility of CrCEST MRI to measure OXPHOS capacity | Baseline
  We will perform CrCEST MRI to map calf muscle Cr recovery kinetics (TCrCEST) following plantar flexion exercise (sec).
To explore feasibility of Fat Fraction MRI to measure OXPHOS capacity | Baseline
  We will perform Dixon MRI to quantify intramuscular fat fraction (IFF %) in the calf.
To explore feasibility of Muscle Ultrasound to measure OXPHOS capacity | Baseline
  Participants will lay supine with legs fully extended with their ankles stabilized in neutral. Customized templates will be strapped on the thigh and consist of five to eight 2-cm slices with a 1-cm gap between slices. Using transmission gel, a continuous, single view will be measured by transversely moving the probe across the thigh in approximately four seconds to acquire images of the rectus femoris (RF) and the vastus lateralis (VL), ensuring minimal pressure is applied to the skin to avoid muscle compression. Bilateral calf muscle CSA will be assessed in the same manner.
To explore feasibility of Muscle Biopsy to measure OXPHOS capacity | Baseline
  A vacuum-assisted biopsy device and ultrasound guidance will be used to obtain skeletal muscle samples. The procedure is performed under local anesthesia with the patient in supine position. The needle will be inserted into the vastus lateralis, accessed through a 2-3 mm incision, under local anesthesia. When the needle is removed, a small section of muscle will remain with the needle. Two samples will be obtained during the procedure. One sample will be analyzed for satellite cell content and morphology. The second sample will be analyzed for mtDNA-CN and epigenetic profile.
To explore feasibility of mtDNA-CN to measure OXPHOS capacity | Baseline
  Peripheral blood samples will be drawn and analyzed for mtDNA-CN, metabolic and epigenetic profile and compared to the muscle sample.

SECONDARY OUTCOMES:
Evaluate muscle strength to measure physical performance | Baseline
  Isokinetic quadricep and ankle strength (Biodex System 4) will be evaluated bilaterally, measured as peak torque (Newton-meters (Nm)) per kilogram (kg) of body weight during cyclical contractions at standard speeds. The average maximum value from each side is used.
Evaluate physical function to measure physical performance | Baseline
  The Timed Up and Go42 captures time to stand, walk 3m, and return to a seated position. The Six Minute Walk tests functional endurance, recorded as the max distance walked 6 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Puneet Bagga, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols